CLINICAL TRIAL: NCT01091779
Title: Changes of Upper and Lower Limb Blood Flow and Vascular Resistance in Hyperbaric Spinal Anesthesia for Transurethral Resection of the Prostate (TURP) Using Duplex Ultrasonography: Comparison of Normotensive and Hypertensive Patients
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2009-0543
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Transurethral Resection of the Prostate (TURP)
Keywords: Male patients scheduled to have spinal anaesthesia for TURP

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypertensive and normotensive

SUMMARY:
Changes of Upper and Lower Limb Blood Flow and Vascular Resistance in Hyperbaric Spinal Anesthesia for TURP Using Duplex Ultrasonography: Comparison of Normotensive and Hypertensive Patients.

ELIGIBILITY:
Inclusion Criteria:

* males (> 65 yr) were scheduled to have spinal anaesthesia for TURP

Exclusion Criteria:

* patients with peripheral vascular disease
* chronic venous insufficiency
* prior deep vein thrombosis (DVT) defined by the presence of thrombosis on duplex or the presence of ultrasonographic signs indicating a previous DVT
* body mass index >35
* prior lower limb surgery due to arterial or venous trauma
* history of diabetes or autonomic deficiency.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Male patients scheduled elective transurethral surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
venous flow velocity, blood volume flow, resistance index, pulsatility index, diameter of popliteal vein | 10 minutes after spinal block

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Kil HK, Suk EH, Lee MH, Bang EC, Hong JY. Venous flow dynamics during spinal block in normotensive and hypertensive elderly patients: a duplex ultrasonographic study. Acta Anaesthesiol Scand. 2012 Mar;56(3):376-81. doi: 10.1111/j.1399-6576.2011.02617.x. Epub 2012 Jan 19. PMID 22260199